CLINICAL TRIAL: NCT06158880
Title: Men's Sexual Risk Behaviors: Alcohol, Sexual Aggression, and Emotional Factors (Extension)
Brief Title: Alcohol & Men's Sexual Risk Behaviors
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Arizona State University (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH); Georgia State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Basic Science
Other Study IDs: STUDY00018369; 4R37AA025212 (NIH)
Record Dates: First submitted 2023-11-28; First posted 2023-12-06 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-07

CONDITIONS: Sexual Behavior; Alcohol Drinking; Sexual Aggression; Emotions
Keywords: Condom use resistance; Emotion dysregulation
MeSH Terms: conditions — Sexual Behavior; Alcohol Drinking | interventions — Alcoholic Beverages

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Alcoholic beverage (Experimental): Participants will receive a dose of alcohol mixed in fruit juice designed to achieve a peak breath alcohol concentration of .08%.
  Interventions: Behavioral: Alcoholic Beverage
- Non-alcoholic beverage (Active Comparator): Participants will receive a beverage that does not contain alcohol (fruit juice only).
  Interventions: Behavioral: Non-alcoholic Beverage
- Partner Negative Mood Manipulation (Experimental): Participants receive an experimental manipulation describing negative emotions in a hypothetical sexual partner.
  Interventions: Behavioral: Partner Negative Mood Manipulation
- Partner Positive Mood Manipulation (Active Comparator): Participants receive an experimental manipulation describing positive emotions in a hypothetical sexual partner.
  Interventions: Behavioral: Partner Positive Mood Manipulation

INTERVENTIONS:
Behavioral: Alcoholic Beverage — Participants will consume an alcoholic beverage (vodka mixed with fruit juice) that is the equivalent of 3-4 standard alcoholic drinks based on their body weight.
  Arms: Alcoholic beverage
Behavioral: Non-alcoholic Beverage — Participants will consume a nonalcoholic beverage (fruit juice) that is the isovolemic equivalent of 3-4 standard alcoholic drinks based on their body weight.
  Arms: Non-alcoholic beverage
Behavioral: Partner Negative Mood Manipulation — Participants will engage in a laboratory task and will then report their own and their partner's emotions following the task.
  Arms: Partner Negative Mood Manipulation
Behavioral: Partner Positive Mood Manipulation — Participants will engage in a laboratory task and will then report their own and their partner's emotions following the task.
  Arms: Partner Positive Mood Manipulation

SUMMARY:
This project extends the investigators' previous research regarding the intersecting risks of alcohol, sexual risk behavior (SRB), and sexual aggression (SA) in male drinkers who have sex with women by examining the mediating and moderating roles of both intrapersonal and interpersonal emotional factors. While independent streams of research consistently document alcohol's role in SRB and SA, the investigators' work has demonstrated that these behaviors are related, and that alcohol exacerbates their likelihood both independently and synergistically. The researchers' investigations focus on a particular type of SRB: men's resistance to condom use with female partners who want to have protected sex. Condom use resistance (CUR) is common and normative among young male drinkers, with up to 80% of men reporting engaging in CUR. Of particular concern, research demonstrates that up to 42% of men report using coercive CUR tactics such as emotional manipulation, deception, condom sabotage, and force to obtain unprotected sex. Investigators will evaluate hypotheses that distal and proximal emotional and alcohol factors influence in-the-moment SRB/CUR intentions as well as daily alcohol use and SRB/CUR. The investigators will also examine whether the relationships among assessed variables are similar across experimental and naturalistic settings. That is, investigate the extent to which men's responses in the lab parallel their real-world drinking and SRB/CUR behaviors, particularly regarding self and partner emotions, empathy, and interpersonal stress.

ELIGIBILITY:
Inclusion Criteria:

* Single
* Male
* Ages 21-30
* Engagement in unprotected intercourse with a woman at least once in the past year
* Consumed alcohol at least 1 time per week in the past 30 days
* Had sex with a woman at least 2 times in the past 30 days

Exclusion Criteria:

* A history of alcohol problems
* A medical condition and/or medications which contraindicate alcohol consumption
* In a relationship that is monogamous and has lasted longer than 6 months

Ages: 21 Years to 30 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Self-defined as male
Enrollment: 320 (Estimated)
Dates: Start 2024-06-17 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Mean score of sexual risk intentions | within one hour of receiving the intervention
  Self-reported ratings of unprotected sex likelihood in a hypothetical scenario Scale range: 1 (not at all likely) to 7 (very likely). A higher value is a worse outcome. This is one total scale (no subscales). Items are averaged to compute a mean score.

SECONDARY OUTCOMES:
Sexual risk behavior | 6 months
  Number of unprotected sexual intercourse events

CONTACTS AND LOCATIONS:
Overall Officials: Kelly Davis, PhD, Principal Investigator — Arizona State University
Locations (1):
- Arizona State University, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: Yes
We will make available individual, de-identified participant data that underlie disseminated results.
Supporting Information: SAP
Time Frame: Immediately following publication and ending 3 years following publication.
Access Criteria: Researchers who provide a methodologically sound proposal for the use of the data. Data will also be made available through the NIAAA Data Archive.